CLINICAL TRIAL: NCT06057675
Title: Subcutaneous Tranexamic Acid in Nasal Mohs Local Flap Reconstruction: Perioperative Bleeding, Edema, and Ecchymosis
Brief Title: Tranexamic Acid in Nasal Mohs Reconstruction
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Priyesh Patel, Asst. Professor of Otolaryngology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 231482
Record Dates: First submitted 2023-09-10; First posted 2023-09-28 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Bleeding; Skin Cancer Face
Keywords: Tranexamic Acid; Mohs Reconstruction
MeSH Terms: conditions — Postoperative Hemorrhage | interventions — Therapeutics; Tranexamic Acid; Lidocaine; Epinephrine; Standard of Care

STUDY DESIGN:
Intervention Model Description: In this study, patients undergoing Mohs reconstruction of the nose with local flap techniques will be randomized to receive either standard of care (subcutaneous injection of local anesthetic, 1% lidocaine with 1:100,000 epinephrine) or TXA treatment (subcutaneous injection of local anesthetic, 1% lidocaine with 1:100,000 epinephrine and TXA 1g/10mL, in 9:1 volume ratio) pre-operatively. Outcomes will include intraoperative bleeding and postoperative swelling and bruising.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient participants will be blinded to the study arm to which they belong. Additionally, the independent reviewer of postoperative photos will be blinded to the study arm to which patients belong. Participation will end at the 7-day follow up appointment, at which time data collection will cease and treatment group will be disclosed to participants.
  Provisions for breaking blinding would include a rare thromboembolic event or anaphylactic event of unknown cause in the immediate postoperative period, or patient desire to terminate involvement in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Active Comparator): The control arm will receive the current standard of care. Before incision, local anesthetic (1% lidocaine with 1:100,000 epinephrine) will be injected subcutaneously into the surgical site. The surgical team will inject approximately 0.8mL per square centimeter of the surgical site area (defect area and undermined tissue area).
  Interventions: Drug: Control (1% lidocaine with 1:100,000 epinephrine)
- Experimental (Experimental): The experimental arm will receive local anesthetic (1% lidocaine with 1:100,000 epinephrine) and TXA (1g/10mL) in a 9:1 volume ratio. This will be injected subcutaneously into the surgical site. The surgical team will inject approximately 0.8mL per square centimeter of the surgical site area (defect area and undermined tissue area).
  Interventions: Drug: Treatment (tranexamic acid and 1% lidocaine with 1:100,000 epinephrine)

INTERVENTIONS:
Drug: Treatment (tranexamic acid and 1% lidocaine with 1:100,000 epinephrine) — Subcutaneous injection of local anesthetic (1% lidocaine with 1:100,000 epinephrine) and tranexamic acid (1g/10mL), mixed in a 9:1 volume ratio.
  Other Names: Tranexamic Acid
  Arms: Experimental
Drug: Control (1% lidocaine with 1:100,000 epinephrine) — Subcutaneous injection of local anesthetic (1% lidocaine with 1:100,000 epinephrine)
  Other Names: Standard of Care
  Arms: Control

SUMMARY:
This study will be a prospective randomized control trial to evaluate the effects of subcutaneously administered TXA among patients undergoing nasal Mohs reconstruction with local flaps at VUMC.

DETAILED DESCRIPTION:
Tranexamic acid (TXA) is an antifibrinolytic agent that acts to decrease bleeding by stabilizing the fibrin matrix involved in the clotting cascade. The use of TXA has been extensively described in the literature to prevent exsanguination in trauma and in various surgical procedures, as well as for heavy menstrual bleeding and epistaxis. Studies have suggested administration of TXA may improve outcomes in aesthetic surgery as well, specifically regarding intraoperative bleeding and postoperative ecchymosis and hematoma formation. TXA may be administered systemically, via IV or PO routes, or locally, via topical application or subcutaneous injection. Local administration allows for similar benefits with minimal risk of systemic effects.

Following facial Mohs reconstruction patients often experience surgical site ecchymosis and swelling, which may be distressing, painful, prolong healing, and result in increased healthcare utilization. Other complications include hematoma, wound dehiscence, and suboptimal scarring. Given the growing body of literature demonstrating the benefits of TXA in surgical bleeding outcomes, TXA may also be beneficial in improving postoperative Mohs complications and patient satisfaction.

To date, no studies have investigated the use of perioperative TXA specifically in nasal Mohs reconstruction. This study will be a prospective randomized control trial to evaluate the effects of subcutaneously administered TXA among patients undergoing nasal Mohs reconstruction with local flaps at VUMC.

ELIGIBILITY:
Inclusion Criteria:

1. Adults at least 18 years of age undergoing local flap reconstruction (bilobe flap, note flap dorsal nasal flap, advancement flap) of a nasal defect following Mohs micrographic surgery. Reconstructive procedures will be performed by Drs. Yang or Patel in the division of Facial Plastic Surgery in the Department of Otolaryngology, Head and Neck Surgery at Vanderbilt University Medical Center.
2. No other facial plastic procedure or sinus surgery performed simultaneously.
3. Lack of all the below exclusion criteria.

Exclusion Criteria:

1. Known allergy to TXA
2. Intracranial bleeding
3. Known defective color vision
4. History of venous or arterial thromboembolism
5. History of coagulation disorder
6. Active thromboembolic disease
7. Severe renal impairment (diagnosis of chronic kidney disease)
8. History of acute myocardial infarction
9. History of stroke
10. History of seizure
11. History of liver failure
12. Preoperative lab results indicating thrombocytopenia (platelets <150,000), increased bleeding risk (PT over 45, INR over 1.2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Surgical site swelling and bruising (surgeon) | One week
  Photos will be taken by a research team member at the first postoperative clinic visit and then analyzed and graded by a blinded reviewer for measures including surgical site bruising and swelling. Surgical site swelling and bruising will be graded on a 4 point scale, with 0 indicating no swelling and bruising and 3 indicating significant swelling and bruising.
Surgical site swelling and bruising (patient) | One week
  Subjective measures of patient perceived swelling and bruising will be collected via a patient completed survey given at the first postoperative clinic visit. Surgical site swelling and bruising will be graded on a 4 point scale, with 0 indicating no swelling and bruising and 3 indicating significant swelling and bruising.
Intraoperative bleeding | Intraoperative
  Intraoperative bleeding will be assessed using the validated Boezaart Bleeding scale (6 point scale, with 0 indicating no bleeding/cadaveric conditions and 5 indicating severe bleeding/constant suctioning required). Values will be assigned by the attending surgeon and recorded by the research team.
Intraoperative bleeding | Intraoperative
  Attending surgeon will score the approximate percent blood saturation of each surgical sponge used in the case. Values from each sponge will be added together for a total cumulative value, with a higher cumulative value indicating a greater amount of intraoperative bleeding.

SECONDARY OUTCOMES:
Postoperative pain | One week
  Subjective measure of patient perceived pain will be collected via a patient completed survey given at the first postoperative clinic visit. Responses will be graded on a 5 point scale, with 1 indicating "no pain" and 5 indicating "severe pain."
Postoperative pain | One week
  Objective measure of pain control will also be collected with an estimate of total amount of opioid pain medication used in the first week after surgery.
Postoperative patient satisfaction | One week
  Subjective measure of postoperative patient satisfaction will be collected via a patient completed survey given at the first postoperative clinic visit. Responses will be graded on a 5 point scale, with 1 indicating "very dissatisfied" and 5 indicating "very satisfied."

CONTACTS AND LOCATIONS:
Overall Officials: Priyesh Patel, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
There are no current plans to make IPD available to other researchers. However, if information is made available, to protect patient privacy, patient names will not be released.